CLINICAL TRIAL: NCT00001291
Title: Investigations of Blood, Synovial Tissue and Synovial Fluids From Patients With Rheumatoid Arthritis and Related Conditions
Brief Title: Genetic and Immune Studies of Rheumatoid Arthritis and Related Conditions
Status: Completed | Type: Observational
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 920065; 92-AR-0065
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-05 (Estimated); Status verified 1999-12

CONDITIONS: Arthritis, Psoriatic; Autoimmune Diseases; Joint Diseases; Osteoarthritis; Rheumatoid Arthritis
Keywords: Osteoarthritis; Psoriatic Arthritis; Rheumatoid Arthritis; Synovial Biopsy; Synovitis; Synovium
MeSH Terms: conditions — Arthritis, Psoriatic; Autoimmune Diseases; Joint Diseases; Osteoarthritis; Arthritis, Rheumatoid; Synovitis

SUMMARY:
This protocol will examine blood, synovial fluid and synovial tissue from patients with rheumatoid arthritis and other chronic inflammatory joint diseases to study genetic and immunologic factors involved in the cause, development and progression of these conditions. Synovial fluid is the lubricating fluid in joints. The synovial membrane is a delicate tissue lining the inner surface of joints, which, in arthritic conditions, thickens and becomes infiltrated with various types of cells.

Patients with rheumatoid arthritis and certain patients with other forms of arthritis may be eligible for this study. Those enrolled will be followed periodically for follow-up and disease evaluation. They may undergo the following procedures:

1. Synovial fluid aspiration, when medically indicated (for example, for joint swelling and inflammation). For this procedure, an area of skin around the joint is numbed with an anesthetic, and a needle is inserted into the joint to withdraw a small fluid sample.
2. Periodic blood sampling, not to exceed 450 milliliters (15 ounces) during any 6-week period, for genetic studies of rheumatoid arthritis. The samples are usually taken at the same times that synovial fluid is withdrawn.
3. Synovial tissues, collected by needle biopsy or during surgical procedures for arthroscopy (examination of the interior of the joint and repair of the joint) or total joint replacement. For the needle biopsy, the skin over the biopsy site is washed and anesthetized. A needle is inserted and fluid is aspirated. The biopsy needle is then inserted through the outer needle and a tissue sample is suctioned.

Patients who qualify for other research studies may be invited to participate.

DETAILED DESCRIPTION:
Blood, synovial fluids and/or synovial tissues will be obtained from patients with rheumatoid arthritis and related chronic inflammatory arthritides. The synovial tissues will be obtained by one of the following methods: a) needle biopsy, or b) at the time of a total joint replacement or a therapeutic arthroscopic procedure. These materials will be utilized for laboratory studies of etiopathogenetic mechanisms of rheumatoid arthritis and related autoimmune joint diseases.

ELIGIBILITY:
Patients with rheumatoid arthritis, particularly new onset disease, but certain patients with other forms of arthritis will also be included.

Significantly swollen or tender knee or significantly swollen shoulders, elbows, wrists, ankles, olecranon bursa or even smaller joints.

Synovial tissue specimens will not be obtained from patients when any of the following conditions are present: abnormal bleeding or clotting tests, platelet count less than 100,000, or sepsis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1991-12; Study Completion 2001-01

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Lafyatis R, Remmers EF, Roberts AB, Yocum DE, Sporn MB, Wilder RL. Anchorage-independent growth of synoviocytes from arthritic and normal joints. Stimulation by exogenous platelet-derived growth factor and inhibition by transforming growth factor-beta and retinoids. J Clin Invest. 1989 Apr;83(4):1267-76. doi: 10.1172/JCI114011. PMID 2784799
- [Background] Kumkumian GK, Lafyatis R, Remmers EF, Case JP, Kim SJ, Wilder RL. Platelet-derived growth factor and IL-1 interactions in rheumatoid arthritis. Regulation of synoviocyte proliferation, prostaglandin production, and collagenase transcription. J Immunol. 1989 Aug 1;143(3):833-7. PMID 2545778
- [Background] Lafyatis R, Thompson NL, Remmers EF, Flanders KC, Roche NS, Kim SJ, Case JP, Sporn MB, Roberts AB, Wilder RL. Transforming growth factor-beta production by synovial tissues from rheumatoid patients and streptococcal cell wall arthritic rats. Studies on secretion by synovial fibroblast-like cells and immunohistologic localization. J Immunol. 1989 Aug 15;143(4):1142-8. PMID 2663990